CLINICAL TRIAL: NCT02379351
Title: Use Of An In-Home Non-Stress Test Device For Remote Fetal Monitoring In A Local High-Risk Obstetric Population
Brief Title: Use Of An In-Home Non-Stress Test Device For Remote Fetal Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 77591
Record Dates: First submitted 2015-02-20; First posted 2015-03-04 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2020-02

CONDITIONS: High Risk Pregnancy
Keywords: Non-stress Test; Fetal Monitoring; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- In-Home Non-Stress Test Device (Experimental): Patients with physician-ordered twice-weekly NSTs scheduled in the OB Diagnostic Center at University of Utah Hospital will be eligible for enrollment. After being taught how to use the Airstrip® Sense4Baby™ system machine, participants will use the device on a weekly basis (at home) until the time of delivery. Participants will also receive an in clinic NST once a week.
  Interventions: Device: In-Home Non-Stress Test Device

INTERVENTIONS:
Device: In-Home Non-Stress Test Device — Airstrip® Sense4Baby™

SUMMARY:
Non-stress tests (NSTs) are used to monitor the health of babies during pregnancy. These tests are currently conducted in clinics and hospitals. This requires travel to a clinic or hospital, sometimes multiple times per week, in order to receive these tests. Technology has been developed that now allows for NSTs to be done in other locations, including home or work. The Airstrip® Sense4Baby™ NST device has been FDA-approved for use by obstetricians in clinical and hospital settings. The investigators are evaluating the use of the Airstrip® Sense4Baby™ NST device in out-of-hospital settings. The investigators would like to know if this type of monitoring is feasible and acceptable to patients and physicians.

DETAILED DESCRIPTION:
Phase I of this study enrolls pregnant women with physician-ordered twice-weekly NSTs scheduled in the OB Diagnostic Center at the University of Utah Hospital. Participants receive an in-clinic NST with the Airstrip® Sense4Baby™ device, are taught how to use the device, and asked to demonstrate their ability to use the device. Once the participant successfully demonstrates use of the monitor the device is given to the participant to use at the scheduled time each week. Patients receive educational materials, including a visuals-enhanced, short quick start guide.

For her remote NST monitoring, the patient will receive a virtual NST appointment. At the time of the scheduled appointment, the patient will apply the monitor and the NST will be read by the mid-level provider staffing the testing center after a thirty-minute strip has been recorded and transmitted to the database. The NST will also be interpreted by the maternal-fetal medicine physician, according to the established workflow. The patient will be notified of the result by a telephone call from the mid-level provider and appropriate follow-up arranged according to the NST management algorithm developed for this study. If the patient has trouble with using the device at home, the patient will be able to talk with the mid-level provider via telephone to troubleshoot issues.

The patient will also continue to receive an NST in clinic weekly. These NST schedules will be repeated on a weekly basis until delivery or until the provider discontinues the NST order.

Patients will be contacted after delivery to assess overall satisfaction with the NST at home versus in clinic.

Phase II of this study will enroll the same patient population (pregnant women with physician-ordered twice-weekly NSTs scheduled). Participants in Phase II may receive NSTs up to twice weekly at home. During regularly scheduled obstetric visits (every 1 to 2 weeks depending on gestational age and circumstances), NSTs will be performed on site. However, we will remove the requirement for once weekly on-site testing at the University of Utah Hospital.

The requirement to be within a 60-mile radius of University Hospital will be removed for Phase II participants. Instead, the requirement will be to be within a 60-mile radius of a hospital with an obstetric unit.

Patients will be contacted after delivery to assess overall satisfaction with the NST at home versus in clinic.

ELIGIBILITY:
Target population: The target population is high-risk pregnant women.

Accessible population: The accessible population is high-risk obstetric patients receiving care throughout the University of Utah Healthcare system and who receive their NSTs at MFDC.

Inclusion Criteria (Phase I):

* Singleton gestation
* Estimated gestational age of 32 0/7 -37 6/7 weeks
* Physician order for twice weekly NSTs
* Live within 60-mile radius of the University of Utah University Hospital
* Reliable access to and connectivity with wireless Internet
* Reliable for communication and follow-up

Exclusion Criteria (Phase I:

* Multifetal gestation
* Maternal age less than 18
* Plans to move prior to end of pregnancy
* No or limited access to internet and/or phone

Inclusion Criteria (Phase II):

* Singleton gestation
* Estimated gestational age of 32 0/7 -37 6/7 weeks
* Physician order for twice weekly NSTs
* Live within 60-mile radius of the University of Utah University Hospital or a hospital with an obstetric inpatient unit
* Reliable access to and connectivity with wireless Internet
* Reliable for communication and follow-up

Exclusion Criteria (Phase II):

* Multifetal gestation
* Maternal age less than 18
* Plans to move prior to end of pregnancy
* No or limited access to internet and/or phone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin AS Clark, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: In-Home Non-Stress Test Device: Patients with physician-ordered twice-weekly NSTs scheduled in the OB Diagnostic Center at University of Utah Hospital will be eligible for enrollment. After being taught how to use the Airstrip® Sense4Baby™ system machine, participants will use the device on a weekly basis (at home) until the time of delivery. Participants will also receive an in clinic NST once a week.
Period: Overall Study
Arm/Group | Experimental: In-Home Non-Stress Test Device
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with physician-ordered twice-weekly NSTs scheduled in the OB Diagnostic Center at University of Utah Hospital
Groups:
- In-Home Non-Stress Test Device: Patients with physician-ordered twice-weekly NSTs scheduled in the OB Diagnostic Center at University of Utah Hospital. Participants utilized the device on a weekly basis (at home) until the time of delivery. Participants also received an in clinic NST once a week.
  In-Home Non-Stress Test Device: Airstrip® Sense4Baby™
Arm/Group | In-Home Non-Stress Test Device
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 31 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Interpretable Results (Participants Who Used the NST Device Correctly)
Description: Number of Interpretable Results (Participants who Used the NST Device Correctly)
Time Frame: Enrollment at 32 0/7 - 37 6/7 weeks gestation through delivery
Population: Patients with physician-ordered twice-weekly NSTs scheduled in the OB Diagnostic Center at University of Utah Hospital. Participants were trained by clinicians at the hospital and then used the device on a weekly basis (at home) until the time of delivery. Participants will also receive an in clinic NST once a week.
Measure: Count of Units; unit: Remote NST's Completed
Units Other Than Participants: Remote NST's Completed
Arm/Group | Experimental: In-Home Non-Stress Test Device
Number analyzed (Participants) | 60
Number analyzed (Remote NST's Completed) | 108
Remote NST's Completed
  Number of Interpretable Results | 107
  Number of Non-Interpretable Results | 1
Statistical Analysis 1: Comparison: Experimental: In-Home Non-Stress Test Device; Test type: Other — This pilot study is primarily descriptive statistics; p = .1, Chi-squared; Data analysis will use mostly descriptive statistics - parametric and nonparametric statistics will be used as indicated (Chi-squared)

2. Secondary Outcome: Provider Satisfaction With Remote NST Compared to On-site NST
Description: Provider Satisfaction With Remote NST Compared to On-site NST
Time Frame: 2 Years
Population: Referring and NST Reading Providers
Measure: Count of Participants; unit: Participants
Groups:
- Providers: Providers involved with NST testing including NST nursing staff, Ordering provider, Interpreting provider.
Arm/Group | Providers
Number analyzed (Participants) | 21
Participants | 21
Statistical Analysis 1: Comparison: Providers; Test type: Non-Inferiority — Likert Scale of Provider Satisfaction; p < 0.01, Chi-squared; Data analysis will use mostly descriptive statistics: parametric and nonparametric statistics will be used as indicated; Likert Scale of Provider Satisfaction

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Experimental: In-Home Non-Stress Test Device
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT02379351/Prot_SAP_000.pdf